CLINICAL TRIAL: NCT03294798
Title: Evaluate the Pharmacokinetic and Pharmacodynamic Profile, Safety, and Tolerability of Escalating Single Dose & Multiple Dose by Using Recombinant Human Serum Albumin/Interferon alpha2b Fusion Protein in Hepatitits B Patients
Brief Title: Study of Recombinant Human Serum Albumin/Interferon alpha2b Fusion Protein in Hepatitis B Patient
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Tianjin SinoBiotech Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 9216-Ib
Record Dates: First submitted 2017-09-21; First posted 2017-09-27 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Hepatitis B Virus
MeSH Terms: conditions — Hepatitis B | interventions — human serum albumin-interferon-alpha-2b fusion protein; peginterferon alfa-2a

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Human Serum Albumin/interferon alpha2b (Experimental): Human Serum Albumin/interferon alpha2b fusion protein 600-900μg,once per two weeks.
  Interventions: Biological: Human Serum Albumin/interferon alpha2b fusion protein
- Pegasys (Active Comparator): Pegasys 180 mcg, once per week
  Interventions: Biological: Pegasys

INTERVENTIONS:
Biological: Human Serum Albumin/interferon alpha2b fusion protein — In experiemental groups, each subject will recieve 600,750,900mg once per two weeks during multiple dose period.
  Arms: Human Serum Albumin/interferon alpha2b
Biological: Pegasys — In comparator group, each subject will recieve 180mcg once per week.
  Arms: Pegasys

SUMMARY:
The purpose of this study is to evaluate the dosages of recombinant human serum albumin/interferon alpha2b fusion protein injection on HBV subjects. The secondary purposes is to get the PK/PD data in recombinant human serum albumin/interferon alpha2b fusion protein injection on HBV subjects.

DETAILED DESCRIPTION:
This is an open-label study that will be conducted at three sites in China to characterize the PK/PD profile, safety and tolerability of Recombinant Human Serum Albumin/interferon alpha2b Fusion Protein in HBV subjects. Subjects will receive a single dose of Recombinant Human Serum Albumin/interferon alpha2b Fusion Protein or active comparator Pegasys at Day 0. A multipule-dose administration in HBV subjects will last 12 weeks after four weeks washout period.

ELIGIBILITY:
Inclusion Criteria:

* HBV patients who have positive HBeAg or HBeAb
* Must be healthy males or females between 18 to 60 years old
* Must have a body mass index (BMI) of 18 to 30 kg/m2
* HBV DNA≥2000 IU/mL
* ALT≥1.3 ULN and ≤10 ULN

Exclusion Criteria:

* Administrated a nucleoside analogues (acid) or interferons against hepatitis B virus drugs, immunosuppressants, immune regulator before 6 months;Or any other against hepatitis b virus therapy at the same time.
* Participated in other clinical trials within a month.
* Allergic to interferon.
* T-Bil ≥2 ULN. ALB<35g/L. PT≥4s.
* Positive HCV-Ab,HEV-Ab,EBV-Ab,CMV-Ab,TPPA,HIV-Ab.
* Organ transplant patients, except cornea or hair transplantation.
* Other hepatopathy exclude NAFLD .
* Drug addiction or alcohol dependence.
* Malignancy(except cured cervical carcinoma in situ, BCC, squamous cell carcinoma) except liver history.
* Serious retinal disease.
* Active hemorrhagic disease or severe hematopoietic dysfunction or blood coagulation disorder.
* Autoimmune disease.
* Uncontrolled diabetes or thyroid disease or beyond grade 2 blood pressure.
* WBC<3×109/L or ANC<1.5 ×109/L or PLT<90 ×109/L or HGB<ULN.
* HCC or AFP>100ng/mL.
* Chronic kidney disease or sCr>ULN.
* Lactating women or pregnancy.
* Cardiovascular and cerebrovascular events within 6 months.
* Neurological or psychiatric disease or family history.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2017-06-13 (Actual); Primary Completion 2019-03-15 (Actual); Study Completion 2021-03-15 (Actual)

PRIMARY OUTCOMES:
the rates of subjects with the level of HBVDNA≤0 IU/mL after treatment | 17 weeks
  HBV DNA

SECONDARY OUTCOMES:
the rates of HBV DNA level decrease by more than 2log10 at the end of 4 weeks and after treatment | 4 weeks and 17 weeks
  HBV DNA
the recovery rates of ALT after treatment | 17 weeks
  ALT
the negative conversion rates of HBsAg/HBeAg and HBeAg seroconversion rates after treatment | 17 weeks
  HBsAg/HBeAg
the rates of HBsAg decrease from baseline after treatment | 17 weeks
  HBsAg

CONTACTS AND LOCATIONS:
Overall Officials: meixia wang, professor, Principal Investigator — Beijing YouAn Hospital; jun li, professor, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University; liang chen, professor, Principal Investigator — Shanghai Public Health Clinical Center
Locations (1):
- Beijing YouAn Hospital, Capital Medical University, Beijing, Beijing Municipality, China